CLINICAL TRIAL: NCT06180265
Title: PRESEPSIN: Biomarker in the Early Diagnosis of Sepsis
Brief Title: The Diagnostic and Prognostic Value of Presepsin in Sepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Foggia (Other)
Responsible Party: Principal Investigator, Cotoia Antonella, Principal Investigator, University of Foggia
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 8/C.E./2020
Record Dates: First submitted 2023-07-25; First posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Septic Shock
Keywords: septic shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- septic shock patients (Other): Septic shock patients undergoing major abdominal surgery treated with polymyxin-B
  Interventions: Diagnostic Test: presepsin, procalciton, endotoxin

INTERVENTIONS:
Diagnostic Test: presepsin, procalciton, endotoxin — measurement of presepsin, procalciton, endotoxin plasmatic levels

SUMMARY:
Intra-abdominal infections are a common cause of sepsis and frequently occur in intensive care unit (ICU) patient. Various markers such as procalcitonin, presepsin and endotoxin are used to identify patients at risk of sepsis or to guide proper treatment.

No studies compared presepsin to procalcitonin and endotoxin in patients treated with by extracorporeal hemoperfusion with a polymyxin-B-adsorbing cartridge (PMX-HA).

DETAILED DESCRIPTION:
Intra-abdominal infections are a common cause of sepsis and frequently occur in intensive care unit (ICU) patient. Various markers such as procalcitonin, presepsin and endotoxin are used to identify patients at risk of sepsis or to guide proper treatment. Particularly, endotoxin can be removed from the blood by extracorporeal hemoperfusion with a polymyxin-B-adsorbing cartridge (PMX-HA).

No studies compared presepsin to procalcitonin and endotoxin in patients treated with PMX-HA. The investigators aim to evaluate the trend and prognostic value of presepsin versus procalcitonin and endotoxin in ICU patients with septic shock from complicated major abdominal surgery, treated with PMX-HA.

ELIGIBILITY:
Inclusion Criteria:

* caucasian patients
* patients undergoing laparoscopic major abdominal surgery

Exclusion Criteria:

* pregnancy,
* organ transplantation,
* palliative care
* metastatic cancer
* head trauma and polytrauma
* coagulopathies
* use of anticoagulants
* neurological disease
* autoimmune disease
* thyroid disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2023-07-19 (Actual)

PRIMARY OUTCOMES:
incidence of mortality at 30-days | up to 30 days
  incidence of mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedali Riuniti, Foggia, Apulia, Italy